CLINICAL TRIAL: NCT07371104
Title: A Multicenter, Open-label, Randomized, Multi-dose, 2-sequence, 2-period, Crossover Bioequivalence Study to Comparison of the Pharmacokinetics and Safety of DWZ2501 and DWC202510 in Patients With Advanced BRCA-mutated High-grade Ovarian Cancer
Brief Title: Bioequivalence Study of DWZ2501 in Patients With Advanced BRCA-mutated High-grade Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWZ2501101
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Ovarian Cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Olaparib, RT) (Experimental): Subjects are randomized into two sequence groups. In Sequence A, subjects receive R then T. T: DWZ2501(Olaparib) R: DW202510(Olaparib)
  Interventions: Drug: DWZ2501 (Olaparib 150mg); Drug: DWC202510 (Olaparib 150mg)
- Sequence B (Olaparib, TR) (Experimental): Subjects are randomized into two sequence groups. In Sequence B, subjects receive T then R.
  T: DWZ2501(Olaparib) R: DW202510(Olaparib)
  Interventions: Drug: DWZ2501 (Olaparib 150mg); Drug: DWC202510 (Olaparib 150mg)

INTERVENTIONS:
Drug: DWZ2501 (Olaparib 150mg) — Subjects receive 600 mg per day, two tablets BID (total 4 tablets), oral administration
Drug: DWC202510 (Olaparib 150mg) — Subjects receive 600 mg per day, two tablets BID (total 4 tablets), oral administration

SUMMARY:
A Multicenter, Open-label, Randomized, Multi-dose, 2-sequence, 2-period, Crossover Bioequivalence Study to Comparison of the Pharmacokinetics and Safety of DWZ2501 and DWC202510 in Patients with Advanced BRCA-mutated High-grade Ovarian Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged 19 years or older at the time of obtaining written informed consent.

2. Patients with advanced high-grade ovarian cancer harboring a BRCA mutation. 3. Subjects who meet at least one of the following criteria:

1. Subjects who have been maintained on an olaparib dosing regimen of 300 mg (two 150 mg tablets) administered orally twice daily for at least 10 consecutive days.
2. Subjects who, in the judgment of the principal investigator require a stable dose of olaparib 300 mg (two 150 mg tablets) administered orally twice daily 4. Subjects with an estimated life expectancy of at least 12 weeks. 5. Subjects with a body mass index(BMI) between 18.50 and 30.00 kg/m² at screening.

Exclusion Criteria:

1. Subjects with a history of hypersensitivity to the investigational product or any of its components.
2. Subjects with any of the following concomitant conditions:

(1) Pneumonitis (2) Myelodysplastic syndrome or acute myeloid leukemia (3) Severe hepatic impairment(Child-Pugh class C). (4) Ongoing active infection or uncontrolled systemic disease (5) Active hepatitis B, hepatitis C, human immunodeficiency virus(HIV) infection, or syphilis.

3. Subjects who have received the following drug and non-drug treatments at screening:

1. Radiotherapy within 4 weeks prior to screening.
2. Other anticancer therapies within 4 weeks prior to screening. 4. Subjects who have undergone major surgery within 4 weeks prior to screening or who have not adequately recovered from a previous major surgery.

5. Subjects who have experienced blood loss of approximately 350 mL or more within 12 weeks prior to screening.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 8, Day 16 after dose administration
  Maximum plasma concentration of olaparib
AUCtau | Day 8, Day 16 after dose administration
  Area under the drug concentration-time curve of olapairb